CLINICAL TRIAL: NCT03179943
Title: GU-114: Overcoming Checkpoint Inhibitor Resistance With Epigenetic Therapy in Urothelial Cancer
Brief Title: Atezolizumab + Guadecitabine in Patients With Checkpoint Inhibitor Refractory or Resistant Urothelial Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Stand Up To Cancer (Other); Van Andel Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-114; SU2C-AACR-CT08-17 (Other Grant/Funding Number: Stand up to Cancer)
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Urothelial Carcinoma
Keywords: bladder cancer; Ureteral Cancer; Urothelial cancer; Urethral cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — atezolizumab; guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Guadecitabine (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Guadecitabine

INTERVENTIONS:
Drug: Atezolizumab — Patients will be administered atezolizumab intravenously on day 1 and day 22 of a 6 week cycle for the period of 8 cycles.
Drug: Guadecitabine — Guadecitabine will be administered subcutaneously on days 1 through 5 of the 6 week cycle for the period of 4 cycles

SUMMARY:
This is a single arm Phase II study with a safety run-in to identify the recommended phase II dose of the combination therapy of atezolizumab and guadecitabine. Patients with recurrent/advanced urothelial carcinoma (stage IV) who had previously progressed on check-point inhibitor therapy with PD-1 or PD-L1 targeting agents are eligible for this study. After a dose that is safe and tolerable has been established, a dose expansion phase (Phase II) will begin. This study will enroll a total of 4 to 53 patients depending upon the number of patients treated in the safety run-in phase and the number of subjects replaced during the phase II portion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed urothelial carcinoma that is advanced or metastatic.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1 and ≥ 1 site safe for biopsy.
3. Patient must agree to provide fresh biopsy specimens and peripheral blood samples at the time of screening and during the study.
4. Patients must have received or be ineligible for platinum based chemotherapy and must have received at least one line of therapy with a PD-L1 or PD-1 targeting agent.
5. Age > 18 years.
6. ECOG performance status ≤ 2
7. Life expectancy ≥ 12 weeks
8. Patients must have normal organ and marrow function as defined below

   * Leukocytes > 3,000/mcL
   * Absolute neutrophil count > 1,500/mcL
   * Platelets > 100,000/mcL
   * Hemoglobin > 9 g/dl (blood transfusion is allowed to meet the eligibility criteria as long as post transfusion hemoglobin is maintained at ≥9.0 g/dL for 7 days or longer)
   * Total bilirubin ≤ 2.5 x institutional upper limit of normal (ULN).
   * AST/ALT (SGOT/SGPT) < 2.5 times institutional normal limits unless liver metastases are present in which case AST and ALT must be ≤ 5 x IULN.
   * Creatinine within normal institutional limits OR
   * Creatinine clearance > 30 Ml/min (Cockcroft-Gault formula or measured with 24h urine)
   * INR or PTT/PT ≤ 1.5 ULN unless patient is on stable therapeutic dose of warfarin
9. Ability to understand and willingness to sign a written informed consent and HIPAA consent document
10. Women of child bearing potential and men must agree to remain abstinent or use adequate contraception (failure rate <1%) for the duration of study and for 90 days after the completion of the therapy.

Exclusion Criteria:

1. Patients who have had anti-cancer therapy within 2 weeks prior to entering the study.
2. Patients receiving any other investigational agents
3. Patients with active or untreated CNS disease. Patients previously treated for CNS disease must be asymptomatic and must not be using steroids for at least 4 weeks prior to starting the study treatment.
4. Patients with active auto-immune disease requiring immunosuppressive medication.
5. Patients treated with systemic immunostimulatory agents (such as interferons, IL 12) within 6 weeks of the start of the treatment or 5 half-lives of the drug, whichever is shorter.
6. Treatment with systemic corticosteroids within 2 weeks prior to the start of the treatment. Patients that require inhaled or low-dose corticosteroids for COPD or asthma, mineralocorticoids are allowed.
7. Patients with active malignancies in addition to urothelial carcinoma.
8. Patients with prior treatment with hypomethylating agents.
9. History of leptomeningeal disease
10. Prior allogeneic stem cell or solid organ transplant.
11. Uncontrolled effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
12. Uncontrolled symptomatic hypercalcemia (>1.5mmol/L ionized calcium or calcium > 12mg/dl or corrected serum calcium > ULN)
13. Mean QT interval corrected for heart rate (QTc) ≥ 470ms calculated from 3 ECGs using Frediricia's correction.
14. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1 except for endocrine AEs managed with replacement therapy. Any other AEs unresolved toxicities grade 2 or more from previous anti-cancer therapy, except alopecia, peripheral neuropathy or non-clinically significant lab abnormalities.
15. Receipt of therapeutic oral or IV antibiotics within 2 weeks prior to the start of the study treatment.
16. Active or prior documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)
17. History of severe allergic, anaphylactic or hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
18. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterations), drug-induced pneumonitis or idiopathic pneumonitis or evidence of interstitial lung disease or active non-infectious pneumonitis.
19. Active tuberculosis
20. Known hypersensitivity to Chinese hamster ovary cell products or any of the study drugs.
21. Administration of a live, attenuated vaccine within 4 weeks of the start of treatment or anticipation that such a live, attenuated vaccine will be required during the study.
22. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
23. Known HIV-positive patients on combination antiretroviral therapy are ineligible.
24. Known history of HBV or HCV infection.
25. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of Guadecitabine in combination of Atezolizumab in safety run-in phase | 2-3 months
  Dose de-escalation study based on standard 3+3 design will be conducted to test two dose levels of guadecitabine: 45mg/m2 and 36mg/m2 to determine MTD
Objective Response Rate (RECIST v 1.1) in Phase II | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years
Progression Free Survival | 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - USC Norris Hospital and Clinics, Los Angeles, California
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No